CLINICAL TRIAL: NCT05003297
Title: Can Neutrophil to Lymphocyte Ratio (NLR) and Platelet to Lymphocyte Ratio (PLR) be Used as Inflammatory Markers to Predict Length of Hospital Stay After Total Laparoscopic Hysterectomy (TLH) for Benign Indications?
Brief Title: Neutrophil to Lymphocyte Ratio (NLR) and Platelet to Lymphocyte Ratio (PLR) as an Inflammatory Markers to Predict Length of Hospital Stay After Total Laparoscopic Hysterectomy (TLH) for Benign Indications
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma ketenci gencer, Dr., Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREHd
Record Dates: First submitted 2021-08-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-07

CONDITIONS: Inflammation; Hospital Stay; Total Laparoscopic Hysterectomy
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients whom were hospitalized for 3 days or less
  Interventions: Other: hemogram inflammatory parameters
- patients hospitalized for more than 3 days
  Interventions: Other: hemogram inflammatory parameters

INTERVENTIONS:
Other: hemogram inflammatory parameters — Neutrophil to Lymphocyte Ratio (NLR) and Platelet to Lymphocyte Ratio (PLR)

SUMMARY:
Due to short hospital stay, rapid return to work, less pain, and good cosmetic results, laparoscopic hysterectomy ( LH) has substantially increased the era of hysterectomy procedures especially for the last two decades. The main reason for this is probably that LH leads to fewer inflammatory responses when compared to open abdominal hysterectomy. Although the inflammatory response is supposed to be lower with total laparoscopic hysteroscopy (TLH), unpredictable inflammatory response as a result of the operation has been still unenlightened and it can be associated with hospital stay.

DETAILED DESCRIPTION:
IInflammatory response after surgery is an ordinary outcome which ends up with tissue repair. The increase in neutrophil levels accompanied with a decrease in lymphocyte levels is characteristic for the inflammatory response. Therefore, neutrophil to lymphocyte ratio (NLR) comes out as a simple index of inflammation. In the literature, NLR was shown not only to be associated with surgical complications but also the length of hospital stays in certain surgeries. Another inflammatory marker index of hemogram is the platelet to lymphocyte ratio (PLR). As a result of endothelial tissue damage, platelets are gathered in the affected area. Therefore, an increase in the number of platelets is inevitable for inflammation. Hence, PLR appears to be another simple index of inflammation due to the increase of platelets and the decrease of lymphocytes. PLR has also shown to be associated with length of hospital stay in various surgeries. NLR and PLR are both newly recommended inflammatory markers to estimate the prognosis of surgical treatment in clinics. Investigations regarding NLR and PLR concerning prognosis of patients after surgeries including gynecological cancer, cardiac surgeries, and emergency surgeries are available in prior literature. Investigators aimed to investigate the possible effects of inflammatory parameters, that can be easily obtained from complete blood count in the post-operative first day of total laparoscopic hysterectomy, to the length of hospital stay in patients without any complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom have undergone TLH

Exclusion Criteria:

* Ureter injury
* Bladder injury,
* Bowel injury,
* Superficial inferior mesenteric artery injury
* Vaginal cuff hematoma
* Vaginal cuff dehiscence
* Endometriosis
* Endometrial cancer
* Cervical cancer
* Chronic lymphocytic leukemia
* Behçet disease
* Electrolyte imbalance
* Thyroid disease
* Using anti-inflammatory medications
* Having severe intraabdominal adhesions

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients whom have undergone TLH without any postoperative surgical complications
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative NLR values compared in patients who were hospitalized for more than 3 days and equal to or less than 3 days. | 4 years
  NLR was calculated by dividing the absolute number of neutrophil to the absolute number of lymphocytes.
Postoperative PLR values compared in patients who were hospitalized for more than 3 days and equal to or less than 3 days. | 4 years
  PLR were calculated by dividing the absolute number of platelets to the absolute number of lymphocytes.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data is available now